CLINICAL TRIAL: NCT06317909
Title: Development of a Novel Non-invasive Inflammometry Following Allergen Challenge in Patients With Mild Allergic Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-03 DONNER-2
Record Dates: First submitted 2024-01-11; First posted 2024-03-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Mild Allergic Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Other): It is an exploratory study. All participants will undergo allergen challenge.
  Interventions: Other: allergen challenge

INTERVENTIONS:
Other: allergen challenge — Patients will undergo inhaled allergen challenge followed by different measures like MRI and induced sputum. At least 4 weeks later patients will undergo segmental allergen challenge followed by different measures like bronchoalveolar lavage.

SUMMARY:
The goal of this exploratory method-development study is to to establish and evaluate novel non-invasive methods to monitor airway inflammation induced by allergen challenge (both by instillation during bronchoscopy and by inhalation) in patients with mild allergic asthma.

The investigator wants to further profile and develop the allergen challenge model by investigating the utility of various non-invasive monitoring methods. The hypothesis of the project is that local inflammatory changes in the lung induced by allergen can be captured by gas-enhanced magnetic resonance imaging (MRI) and analysis of exhaled breath.

The validation of cellular outcome measures and non-invasive inflammometry can be used in future clinical trials for proof of concept of novel anti-inflammatory medications.

Participants will undergo

* methacholine challenge
* 2 inhaled allergen challenges
* 2 MRI with hyperpolarized xenon and gadolinium based contrast agent
* 2 bronchoscopies with bronchoalveolar lavage (BAL)
* segmental allergen challenge during the first bronchoscopy
* spirometry
* skin prick test and skin prick dilution tests
* measurement of particles in exhaled air
* nasal filter
* nasal lavage
* sputum induction
* peak flow meter tests
* exhaled NO (nictric oxide)
* blood sampling (in total approx. 190 ml)

DETAILED DESCRIPTION:
An individual study participation takes about 6 to 8 weeks for the experimental phase not including a screening phase that can add up to 8 weeks. The study consists of 10 visits. All visits take place at Fraunhofer ITEM in Hannover.

During screening an inhaled allergen challenge will be performed to decide about eligibility. During the experimental part another inhaled allergen challenge, 2 magnetic resonance imaging (MRI) and 2 bronchoscopies with segmental allergen challenge will be performed.

Methacholine Challenge:

The methacholine bronchial challenge will be performed in accordance with study sites Standard Operating Procedure (SOP). Methacholine will be used according to the manufacturers' instruction. After an initial saline inhalation as a reference, the percent decrease in Forced Expiratory Volume in the first second (FEV1) after each succeeding concentration of methacholine will be determined until the FEV1 drops to 80% of the reference value. An interpolated PC20 (aerosol concentration of methacholine leading to a 20% fall in the FEV1) will be calculated.

Inhaled allergen challenge:

For the inhaled allergen challenge the allergen most likely to induce allergic airway responses will be selected during the screening period. The allergens used for provocation in this study will be lyophilized allergen extracts of respective allergen (LETI Laboratories) developed and licensed for provocation testing.

The starting concentration of allergen extract to be given by inhalation will be calculated based on the prick dilution test as well as the methacholine challenge in order to obtain the allergen concentration that is predicted to cause a 20% decrease in FEV1 ( PC20).

Bronchoscopies with BAL and segmental allergen challenge:

Bronchoscopy will be performed according to the study sites which is consistent with international recommendations for fiberoptic bronchoscopy. In this clinical investigation, two bronchoscopies will be conducted under identical conditions 24 hours apart. Before instillation of allergen, a baseline lavage will be performed during the first bronchoscopy. . Thereafter, a control challenge will be performed by injecting 10 ml of 37°C sterile 0.9% saline.During the second bronchoscopy after 24 hours, BAL from the two challenged segments will be collected. The allergen used for inhaled provocation will be used for segmental provocation as well.

Magnetic resonance imaging:

MRI will be performed at the Clinical Research Center by the Institute for Radiology using a Siemens Avanto 1.5T scanner. In order to assess local inflammation by proton MRI, various sequences will be applied during the imaging session. In addition, gas-enhanced protocols with hyperpolarized xenon will be applied according to the study sites SOP. For the assessment of pulmonary perfusion, a gadolinium based contrast agent (Gadopentetat - Dimeglumin) will be given iv during each MRI scan. It will be 1/3 of the regular dose for this contrast agent.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Male and female subjects aged 18-65 years. Women will be considered for inclusion if they are:

   * Not pregnant, as confirmed by pregnancy test (see assessment schedule), and not nursing.
   * Of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre-menarcheal or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the Screening Visit).
   * Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence, implants, injectables, combined oral contraceptives, hormonal Intrauterine Devices (IUDs) or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
3. History of mild asthma for at least 12 months prior to the Screening Visit that is well controlled with Short Acting Beta-Adrenergic Stimulator (SABA) only.
4. Body mass index between 18 and 32 kg/m2
5. Normal pulmonary function with forced Expiratory Volume in the first second (FEV1) ≥80% of predicted normal and FEV1/Forced Vital Capacity(FVC) ≥70% at Screening Visit. Calculations will be based on Global Lung Function Initiative (GLI) formula. If the participant fails to meet this criterion on the first measurement, spirometry may be repeated twice.
6. Positive skin prick test (wheal diameter reaction ≥3 mm) for the respective challenge aeroallergen (i.e. tree, weed, grass or house dust mite) at or within 12 months prior to the Screening Visit (if performed and documented at Fraunhofer ITEM).
7. Positive early and late asthmatic response upon incremental inhaled allergen challenge at or prior to the Screening Visit (if performed and documented at Fraunhofer ITEM).
8. Production of adequate sputum with ≥1 x 106 total non-squamous cells at or within 12 month prior to the Screening Visit 1 (if not performed and documented at Fraunhofer ITEM).
9. Nonsmokers with a history of less than 1 pack year having been nonsmokers for at least one year.

Exclusion Criteria:

1. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, lung function or ECG at Screening Visit, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study.
2. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, metabolic disease (asymptomatic Gilbert's syndrome is allowed), endocrine disease (stable and asymptomatic hypothyroidism with or without hormone replacement therapy (HRT) is allowed), or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
3. Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for pain relief, contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements.
4. Specific Immunotherapy (SIT) within three years prior to the study.
5. Intake of systemic or inhaled steroids within 4 weeks before Screening Visit 1a.
6. Respiratory tract infection (RTI) within 4 weeks before Screening Visit 1a.
7. Mild to moderate asthma exacerbation within 3 months before Screening Visit 1a.
8. Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
9. Suspected hypersensitivity to any ingredients of the medication in line with bronchoscopy (bronchodilators, sedatives and local anesthetics).
10. Conditions or factors, which would make the subject unlikely to be able to undergo bronchoscopy or allergen challenge.
11. Conditions or factors, which would make the subject unlikely to undergo MRI (e.g. due to claustrophobia, cardiac pacemaker, hypersensitivity to MR i.v. contrast imaging agents).
12. Participation in another clinical trial with Investigational Medicinal Product (IMP) 30 days or 5 half-lives, whichever is longer, prior to enrollment.
13. Participation in the observation period of a competing study within 30 days prior to Screening.
14. Segmental allergen challenge three months prior to bronchoscopy.
15. Donation of more than 400 ml of blood the preceding 60 days before screening.
16. History of regular drug or alcohol abuse
17. Risk of non-compliance with study procedures.
18. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Exploratory (1. priority) Changes in soluble mediators [i.e. IL-4, IL-5, IL-8, IL-13, IL-33, TSLP, IL-1, IL-6, INF-alpha, MMP-9, CXCL1, SP-D, albumin] in Bronchoalveolar lavage (BAL) after segmental allergen challenge | 24 hours after segmental allergen challenge
  Quantification of allergic inflammatory response induced by segmental allergen challenge in BAL by analyzing soluble mediators using Meso Scale Discovery (MSD) multiplex assays -> At least, but not limited to Interleukin(IL)-4, IL-5, IL-8, IL-13, IL-33, Thymus-Stroma-Lymphopoietin (TSLP), IL-1, IL-6, Interferon-alpha (INF-alpha), Matrix-Metallopeptidase 9 (MMP-9), Chemokine (C-X-C motif) ligand 1 (CXCL1), Surfactant protein D (SP-D), albumin [pg/ml]
Exploratory (1. priority) Changes in soluble mediators [i.e. IL-4, IL-5, IL-8, IL-13, IL-33, TSLP, IL-1, IL-6, NF-alpha, MMP-9, CXCL1, SP-D, albumin] in Sputum after inhalative allergen challenge | 24 hours after segmental allergen challenge
  Quantification of allergic inflammatory response induced by inhalation in sputum by analyzing soluble mediators using MSD multiplex assays -> At least, but not limited to IL-4, IL-5, IL-8, IL-13, IL-33, TSLP, IL-1, IL-6, NF-alpha, MMP-9, CXCL1, SP-D, albumin [pg/ml]
Exploratory (1. priority) Changes in non-invasive exhaled particles [i.e.IL-4, IL-5, IL-8, IL-13, IL-33, TSLP, IL-1, IL-6, NF-alpha, MMP-9, CXCL1, SP-D, albumin]after inhalative allergen challenge | before, 3, 6 and 24 hours after inhaled allergen challenge
  Quantification of allergic inflammatory response induced by inhalation in non-invasive exhaled particles at multiple time-points by analyzing soluble mediators using MSD multiplex assays -> At least, but not limited to IL-4, IL-5, IL-8, IL-13, IL-33, TSLP, IL-1, IL-6, INF-alpha, MMP-9, CXCL1, SP-D, albumin [pg/ml]
Exploratory (1. priority) Changes in non-invasive exhaled particles [i.e.IL-4, IL-5, IL-8, IL-13, IL-33, TSLP, IL-1, IL-6, NF-alpha, MMP-9, CXCL1, SP-D, albumin]after segmental allergen challenge | before, 3, 6 and 24 hours after segmental allergen challenge
  Quantification of allergic inflammatory response induced by segmental allergen challenge in non-invasive exhaled particles at multiple time-points by analyzing soluble mediators using MSD multiplex assays -> At least, but not limited to IL-4, IL-5, IL-8, IL-13, IL-33, TSLP, IL-1, IL-6, INF-alpha, MMP-9, CXCL1, SP-D, albumin [pg/ml]
Exploratory (1. priority) Changes in cell analyzation in BAL [i.e.total cells, neutrophil granulocytes, eosinophil granulocytes, basophil granulocytes, monocytes/macrophages, lymphocytes and dendritic cells] after segmental allergen challenge | 24 hours after segemental allergen challenge
  Quantification of allergic inflammatory response induced by segmental allergen challenge in BAL by analyzing cellularity and functionality using microscopy, flow cytometry and chipcytometry ->At least, but not limited to total cells, neutrophil granulocytes, eosinophil granulocytes, basophil granulocytes, monocytes/macrophages, lymphocytes and dendritic cells [×10^6 cells/ml]
Exploratory (1. priority) Changes in cell analyzation in Sputum [i.e.total cells, neutrophil granulocytes, eosinophil granulocytes, basophil granulocytes, monocytes/macrophages, lymphocytes and dendritic cells] after inhalative allergen challenge | before, 6 and 24 hours after inhaled allergen challenge
  Quantification of allergic inflammatory response induced by inhalation in sputum by analyzing cellularity and functionality using microscopy, flow cytometry and chipcytometry -> At least, but not limited to total cells, neutrophil granulocytes, eosinophil granulocytes, basophil granulocytes, monocytes/macrophages, lymphocytes and dendritic cells [×10^6 cells/ml]

SECONDARY OUTCOMES:
Exploratory (2. priority) Detection of Ribonucleic acid (RNA) in exhaled particles | before, 3, 6, and 24 hours after allergen challenge
  Detection of RNA in exhaled particles ->Verification and quantification of RNA
Exploratory (2. priority) Changes in Fractional exhaled nitric oxide (FeNO) after inhalative allergen challenge | before, 3, 6, and 24 hours after inhaled allergen challenge
  Quantification of inflammation in the central airways by FeNO in the kinetic of the allergic response after inhalation challenge -> Measurement of FeNO [ppB] and comparison with induced sputum
Exploratory (2. priority) Changes in FeNO after segmental allergen challenge | before, 3, 6 and 24 hours after segmental allergen challenge
  Quantification of inflammation in the central airways by FeNO in the kinetic of the allergic response after segmental challenge -> Measurement of FeNO [ppB] and comparison with induced sputum
Exploratory (2. priority) Quantification of regional ventilation, perfusion, and diffusion by magnetic resonance imaging (MRI) | before and 6 hours after inhaled allergen challenge
  Quantification of regional ventilation, perfusion, and diffusion assessed by MRI
  -> change from baseline of MRI assessed parameters in relation to inflammatory reaction (eosinophil numbers [×10^6 cells/ml] in sputum and BAL) and pulmonary function (FEV1 and maximal forced expiratory flow (MFEF) of 25 to 75% of Vital Capacity of the lungs (MFEF25-75))

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No